CLINICAL TRIAL: NCT06919874
Title: Dyadic Yoga Program for Patients Undergoing Thoracic Radiotherapy and Their Family Caregivers: The Testing of a Mobile Application Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0128; NCI-2025-02119 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thinking Out Loud Group (Experimental): Participants will be identified using the electronic clinic appointment systems for the thoracic radiation clinic and prescreened for their date of birth (i.e. minimum 18 years old), disease, treatment schedule, ECOG and other criteria (e.g., exercise intolerance, cognitive deficits).
  Interventions: Behavioral: Thinking out Loud Session

INTERVENTIONS:
Behavioral: Thinking out Loud Session — Participants will complete one thinking out loud session (approx. 60 minutes). The session will be led by a yoga therapist (see below) either in person at the hospital or via Zoom. Individual patients, caregivers or patient-caregiver dyads will attend the session. Each participant will need to either bring their own device or will use an institutional loaner device if no personal device is available. During the session, participants will be asked to download the app from the device appropriate app store and open the app. Then, we will implement the thinking out loud methods asking participants to continuously think out loud, meaning verbalizing their thoughts as they move through the user interface of the app. The sessions will be audio recorded with permission obtained during the consent process. Specific feedback will be requested using a semi-structured interview approach

SUMMARY:
The goal of the trial is to test the usability, feasibility and acceptability of an unsupervised, appbased yoga program for participants undergoing thoracic RT and their caregivers.

DETAILED DESCRIPTION:
Primary Objective:

The Investigators propose to test the usability, feasibility and acceptability of an unsupervised, app-basedyoga program for patients undergoing thoracic RT and their caregivers. The Investigators specific aims will be carried out in two parts:

Part 1:

• The Investigators will perform the initial usability testing of the working prototypes of both iOS and Android versions to determine whether users can complete the required tasks successfully and independently and to identify problems with navigation and functioning.

The Investigators primary objective is to:

Aim 1: Finalize the working prototype of the yoga app using the feedback of 10 participants-caregiver dyads (mixed-methods study).

Part 2:

• The Investigators will measure feasibility (e.g., consent and retention rates, adherence), usability of the app, and acceptability of the app-based program in 20 newly recruited participants-caregiver dyads. As an exploratory outcome, the investigators include pre- and post-intervention assessments of objective physical function and self-reported QOL. The Investigators will also complete semi-structured interviews to collect qualitative data on participants' evaluation of the mobile app and their experience in participating in this research.

Specific aims are:

Aim 1: Examine the feasibility, usability, and acceptability of an app-based yoga program in 20 patient-caregiver dyads (single-arm trial).

Aim 2: Understand the trial participants' experiences with the mobile app delivery including suggestions for improvement using qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with a non-small cell lung cancer or esophageal cancer and going to receive at least 24 fractions thoracic RT
2. Have an ECOG performance status of <2
3. Have a family caregiver (e.g., spouse, sibling, adult child) willing to participate

Both patient and caregiver must meet all the following criteria:

1. Be >18 years old
2. Be able to read and speak English
3. Be able to provide informed consent
4. Have regular (self-defined) access to Wi-Fi/High speed internet access

Exclusion Criteria:

1. Experiences cognitive deficits that would impede the completion of self-report instruments as deemed by their attending oncologist
2. Experiences contraindications to exercise as determined by the clinical team
3. Regularly (self-defined) participants in a yoga program in the year prior to diagnosis

Participants who participated in part 1 are ineligible to participate in part 2 of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, MA,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org